CLINICAL TRIAL: NCT04845100
Title: The Effect of Animal Assisted Activities on the Stress and Social Anxiety Levels of Disabled Children
Brief Title: Animal Assisted Activities on the Stress and Social Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Şeyma Demiralay (Other)
Responsible Party: Sponsor-Investigator, Şeyma Demiralay, Graduate student, Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 013
Record Dates: First submitted 2021-01-19; First posted 2021-04-14 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Stress; Social Anxiety; Disabling Disease; Animal Communication; Nursing Caries; Child
Keywords: pet therapy; disabled child; stress; social anxiety
MeSH Terms: conditions — Animal Communication

STUDY DESIGN:
Intervention Model Description: The study is a single blind randomized controlled study designed in a pretest, posttest and follow-up design.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The Effect Of Animal Assisted Activities On The Stress And Social Anxiety Levels Of Disabled Children
  Animal Assisted Activity Program (HayDAP)
  Interventions: Other: Animal Assisted Activity Program
- Control group (Other): No intervention
  Interventions: Other: Animal Assisted Activity Program

INTERVENTIONS:
Other: Animal Assisted Activity Program — Animal Assisted Activity Program (HayDAP)
  1. st week (Pre-test, introduction-introduction)
  2. nd week (Information about cats)
  3. th (Cat story reading)
  4. th week (Teaching songs, poems, rhymes about cat)
  5. th week (Making / decorating a cat house)
  6. th week (Participation in the rehabilitation program with the treatment animal)
  7. th week (Evaluation and closing, last test)

SUMMARY:
ABSTRACT Objective: The aim of the study is to determine the effects of animal-assisted activities on the stress and social anxiety levels of physically disabled children.

Method: The research was carried out in two separate Special Education and Rehabilitation Centers providing education under the Antalya Provincial Directorate of National Education. The data of the study were obtained between November 2019-September 2020. The study is a single blind randomized controlled study designed in a pretest, posttest and follow-up design. The study was carried out in two different institutions to prevent contamination. Institutions are determined by an independent lottery method. The sample of the study consisted of 44 physically disabled children between the ages of 8-11, as the intervention group (n: 21) and the control group (n: 23). A 45-60 minute structured animal supported activity program (HayDAP) was applied to the intervention group, once a week for 7 weeks. Interviews were conducted individually. The data of the study were obtained using Personal Information Form (KBF), Perceived Stress Scale (PSS) and Social Anxiety Scale for Children. Follow-up evaluation was made at the end of the 1st month following the completion of the application. There was no intervention in the control group. The data were analyzed using the Pearson Ki-Square Test in SPSS 23.0 package program, Fisher's Exact Test if large, Shapiro-Wilks Test, Box M, Bonferroni and mixed pattern ANOVA tests. A 95% significance level (or α = 0.05 margin of error) was used to determine the differences in the analyzes.

DETAILED DESCRIPTION:
ANIMAL ASSISTED ACTIVITY PROGRAM (HayDAP):

1. st week (Pre-test, introduction-introduction) Goal. Developing a trusting relationship
2. nd week (Information about cats) Purpose: To strengthen the bond that develops between the child and the application animal
3. th (Cat story reading) Purpose: To evaluate the emotions and solutions in the face of stressful life events in the face of the story.
4. th week (Teaching songs, poems, rhymes about cat) Objective: To determine the factors that may cause social anxiety and to support the increase of self-confidence in the child.
5. th week (Making / decorating a cat house) Purpose: Discussing the roles and relationships of the child in his / her social environment and developing awareness with examples of cats.

   Improving communication and problem solving skills
6. th week (Participation in the rehabilitation program with the treatment animal) Purpose: To monitor the child's adherence to treatment Evaluating the child's compliance with the treatment during physiotherapy activities while being observed by the application cat and the practitioner
7. th week (Evaluation and closing, last test) Purpose: Finishing the whole process by passing A healthy termination of the bond formed with the practice cat

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* Being in the age range of 8-11,
* Only being physically disabled,
* Reading and writing,
* Parent's consent for the child to participate in the study

Exclusion Criteria:

* Do not have an obstacle about the message
* Being in any chronic disease with immune deficiency,
* Don't have any animal allergies,
* Application being afraid of animals,
* Have an existing animal of your own, past or present

Extraction Criteria:

* Not participating in the interview for more than 2 weeks,
* Development of a medical condition that prevents communication,
* Participant's right to withdraw from the research in line with his family or his own request

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Stress | 7 Weeks, 1 Month
  Perceived Stress Levell Scale; This one-dimensional scale consists of 9 items. It has a 4-point Likert type rating.
  The scores that can be obtained from the scale are between 9 and 36.
  The high scores on the scale questions indicate that the individual's stress level is means to be high.

SECONDARY OUTCOMES:
Social Anxiety | 7 Weeks, 1 Month
  Social Anxiety Scale for Children-Revised; This one-dimensional scale has a 5-point Likert-type scale consisting of 18 items.
  The scores that can be obtained from the scale are between 18 and 90.
  The higher the score, the higher the social anxiety level.
Blood Pressure | Only intervention group, every pre-intervention and post-intervention: During HayDAP intervention, for 7 weeks, before and after each application
  Blodd Pressure

CONTACTS AND LOCATIONS:
Overall Officials: İlkay KESER, Ass. Prof., Study Director — Akdeniz University
Locations (1):
- Şeyma Demiralay, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Animal Assisted Activity Program (HayDAP)
  1. st week (Pre-test, introduction-introduction)
  2. nd week (Information about cats)
  3. th (Cat story reading)
  4. th week (Teaching songs, poems, rhymes about cat)
  5. th week (Making / decorating a cat house)
  6. th week (Participation in the rehabilitation program with the treatment animal)
  7. th week (Evaluation and closing, last test)